CLINICAL TRIAL: NCT05358301
Title: Novel Strategies for Obesity Prevention and Management With the Probiotic Lactiplantibacillus Plantarum IMC 510 (PRO-Weight-Control Study)
Brief Title: Targeting Obesity With the Probiotic Lactiplantibacillus Plantarum IMC 510 (PRO-Weight-Control Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Francesco Sofi, Associate Professor of Clinical Nutrition, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO-Weight-Control
Record Dates: First submitted 2022-03-21; First posted 2022-05-03 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Obesity
Keywords: obesity; probiotic; Lactiplantibacillus Plantarum; gut microbiota; clinical trial
MeSH Terms: conditions — Obesity | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized double-blind parallel controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: By keeping both the experimenters and the participants blind, bias is less likely to influence the results of the experiment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Probiotic food supplement produced by SYNBIOTEC S.r.l.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo food supplement.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic food supplement produced by SYNBIOTEC S.r.l. Each capsule of SYNBIO®slim contains the probiotic strain Lactiplantibacillus Plantarum IMC 510 at a concentration of 15 billion live cells (CFU/capsule). The assumption is of n°1 capsule/day, preferably at breakfast, for 3 months. The capsules can be opened and their content can be dispersed in a cold liquid or at intake temperature or in semi-solid food. Always store in original container or in a clean covered container, out of the reach of children. When stored in a dry, clean environment, out of direct sunlight, the product has a shelf-life of at least 24 months. Samples of probiotic supplement in closed and sealed boxes will be provided to subjects participating at the beginning of the study, in quantities sufficient for the entire duration of the study (90 capsules for 3 months).
  Arms: Probiotic
Dietary Supplement: Placebo — N°1 capsule/day of placebo food supplement (i.e., capsules without added probiotics), with the same intake modalities as probiotic.
  Arms: Placebo

SUMMARY:
In recent decades, the prevalence of obesity has reached epidemic proportions, with the number of overweight or obese individuals continuing to increase worldwide. Advances in recent research have allowed a better characterization of the etiology of obesity, demonstrating the involvement of the gut microbiota. In fact, while signals from the brain influence gut function, the gut microbiota has been shown to modulate brain functions involved in the regulation of stress, depression and anxiety, which are closely linked to obesity. Oral administration of probiotics has been proposed as a valid way to modulate the gut ecosystem to promote weight reduction. Preliminary data showed that obese rats treated with probiotics containing the probiotic strain Lactiplantibacillus Plantarum IMC 510 exhibited significantly lower weight and food intake than untreated obese rats. Although exercise and diet are the first lines of intervention to be recommended, there are often failures or poor outcomes. There is currently increased interest in alternative and effective shorter-term, non-pharmacological approaches to weight control that involve the use of natural active ingredients. Thus, the aim of this intervention study is to investigate whether a probiotic supplementation with Lactiplantibacillus Plantarum IMC 510 could be beneficial for the weight reduction of people with obesity.

DETAILED DESCRIPTION:
Background

Obesity is a multifactorial disease characterized by a chronic imbalance between energy intake and energy expenditure. Risk factors for weight excess are genetic, metabolic, hormonal, psychological, and social, as well as factors related to diet, sedentary lifestyle, and medication intake. Obesity is associated with an increased risk of onset of several metabolic diseases (high blood pressure, dyslipidemia, diabetes mellitus, metabolic syndrome), cardiovascular diseases (cerebral strokes, myocardial infarction), gastrointestinal diseases (esophageal reflux, cholelithiasis, pancreatitis, hepatopathy), respiratory diseases (apnea, respiratory failure), cancer (higher incidence of cancer and worsening of prognosis), osteoarticular diseases (osteoporosis, osteoarthritis), psychological diseases (depression, low self-esteem, relationship problems).

In recent decades, the prevalence of obesity has reached epidemic proportions. In fact, current data estimate that approximately 600 million people worldwide are obese, with an additional 1.9 billion overweight. Moreover, recent trend analyses show that the number of individuals who are overweight or obese continues to increase worldwide.

Advances in recent research have allowed for better characterization of the etiology of obesity, highlighting the potential contribution of factors not traditionally considered to be involved in changes in energy balance and body composition. Experimental and clinical studies have also demonstrated the role of the gut microbiota in the regulation of energy balance and the occurrence of excess body weight. In this regard, it has been suggested that lean and obese human subjects differ in the composition of their gut microbiota, and that probiotics and prebiotics can be used to modify the microbiota to prevent body weight gain. The bidirectional gut-brain connection allows signals from the brain to influence motility, appetite sensations, secretions, and permeability of the gut. Studies have demonstrated the role and importance of the gut microbiota in modulating central nervous system activity, so some gut messages may influence brain functions involved in the regulation of stress, depression, and anxiety, which are closely related to obesity. Consequently, the gut microbiota is a potential modifiable target for the prevention and/or treatment of obesity. In fact, the gut microbiota has recently been shown to play a complex role in body weight regulation and some probiotic strains have been able to ameliorate obesity status and related metabolic disorders. Preliminary data showed that obese rats treated with probiotics containing the probiotic strain Lactiplantibacillus Plantarum IMC 510 exhibited significantly lower weight and food intake than untreated obese rats.

Oral administration of probiotics has been proposed as a viable way to modulate/modify the gut ecosystem to promote weight reduction; however, the mechanisms by which probiotic supplementation may affect the gut microbiota of obese individuals are largely unknown. In addition, byproducts of the bacterial fermentation process may also reduce appetite and increase feelings of satiety, and through modulation of bile acid metabolism, the microbiota may reduce diet-induced obesity through increased energy expenditure. In addition, gut bacteria can manipulate an individual's taste and food preferences.

Over the past 25 years, more than 120 drugs have been studied for the treatment of obesity, but only very few have been approved and maintained on the market. Although exercise and diet are the first lines of intervention in correcting overweight, obesity and related metabolic diseases, because they are measures that must be adopted and followed for a long period of time, often experience failure or poor outcomes. Currently there is an increased interest in alternative and effective short term non-pharmacological approaches to weight control that involve the use of natural active ingredients. The use of specific probiotics could represent the future weapon to fight obesity through the modulation of the intestinal microbiota, which is becoming more and more important as a critical point both for the appearance of many diseases (if altered) and for the possibility of curing them by intervening to restore the intestinal flora.

Objectives of the study

The present clinical study is directed to the evaluation of the efficacy of a probiotic formulation containing the probiotic strain Lactiplantibacillus Plantarum IMC 510 in inducing and supporting weight loss and reduction of body circumferences in overweight or obese subjects through the regularization of appetite with consequent reduction of food intake.

Primary Objectives:

1) To evaluate weight reduction in obese and/or overweight subjects after 3 months of treatment with probiotic or placebo.

Secondary Objectives:

1. Collection of blood and fecal samples at recruitment, after 3 months of treatment (probiotic or placebo), and after a 1-month final wash out.
2. Measurement of BMI, body circumferences, body composition such as fat mass, lean mass, after 3 months of probiotic or placebo treatment, and after 1 month of wash out
3. Evaluation of general well-being, eating habits and any gastrointestinal symptoms
4. Comparison of hematological and biochemical parameters related to obesity at baseline, after 3 months of probiotic or placebo intervention, and after 1 month of washout
5. Analysis of the composition of the intestinal microbiota and the production of short-chain fatty acids (SCFA) and bile acids (FBA).

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-65 years of age
* Obesity (BMI >30 kg/m2, class I, II, III) and overweight (BMI 25-29.9 kg/m2)
* Willingness to cooperate during the study and ability to follow guidelines
* Willingness to complete questionnaires and diaries associated with the study and to complete all clinical visits
* Willingness to discontinue functional foods and dietary supplements with probiotics, laxatives and body weight control substances
* Ability to provide informed consent

Exclusion Criteria:

* Continued use of probiotics in the two months prior to treatment
* Use of other treatments (medications or nutritional programs) that affect body weight, food intake and/or energy expenditure
* Postmenopausal women
* Pregnant or lactating
* Enrolled in another obesity treatment program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Body weight | 2 months
  Changes of body weight from baseline assessed through a balance

SECONDARY OUTCOMES:
Fat mass | 2 months
  Changes of fat mass from baseline assessed through a bioelectrical impedance analysis device (BIA Akern, 101 Sport Edition).
Fat-free mass | 2 months
  Changes of fat-free mass from baseline assessed through a bioelectrical impedance analysis device (BIA Akern, 101 Sport Edition).
Total body water | 2 months
  Changes of total body water from baseline assessed through a bioelectrical impedance analysis device (BIA Akern, 101 Sport Edition).
White blood cells | 2 months
  Changes of white blood cells from baseline assessed to standard laboratory procedures.
Red blood cells | 2 months
  Changes of red blood cells from baseline assessed to standard laboratory procedures.
Hemoglobin | 2 months
  Changes of hemoglobin from baseline assessed to standard laboratory procedures.
Glucose | 2 months
  Changes of glucose from baseline assessed to standard laboratory procedures.
Urea | 2 months
  Changes of urea from baseline assessed to standard laboratory procedures.
Creatinine | 2 months
  Changes of creatinine from baseline assessed to standard laboratory procedures.
Sodium | 2 months
  Changes of sodium from baseline assessed to standard laboratory procedures.
Potassium | 2 months
  Changes of potassium from baseline assessed to standard laboratory procedures.
Calcium | 2 months
  Changes of calcium from baseline assessed to standard laboratory procedures.
Magnesium | 2 months
  Changes of magnesium from baseline assessed to standard laboratory procedures.
AST | 2 months
  Changes of AST from baseline assessed to standard laboratory procedures.
ALT | 2 months
  Changes of ALT from baseline assessed to standard laboratory procedures.
Triglycerides | 2 months
  Changes of triglycerides from baseline assessed to standard laboratory procedures.
Total cholesterol | 2 months
  Changes of total cholesterol from baseline assessed to standard laboratory procedures.
HDL-cholesterol | 2 months
  Changes of HDL-cholesterol from baseline assessed to standard laboratory procedures.
LDL-cholesterol | 2 months
  Changes of LDL-cholesterol from baseline assessed to standard laboratory procedures.
Uric Acid | 2 months
  Changes of uric acid from baseline assessed to standard laboratory procedures.
eGFR | 2 months
  Changes of eGFR from baseline assessed to standard laboratory procedures.
Gastrointestinal and systemic symptoms | 2 months
  Changes of gastrointestinal and systemic symptoms from baseline assessed through a modified form of the Global Assessment of Improvement Scale (GAI), with a total score ranging from 0 to 56, with higher scores meaning an improvement of the symptoms and the Symptom Severity Scale (SSS), with a total score ranging from 0 to 500, with higher scores meaning more severe symptoms.
Gut microbiota | 2 months
  Changes of gut microbiota from baseline assessed by Illumina MiSeq platform.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Sofi, Prof., Principal Investigator — Unit of Clinical Nutrition, University hospital of Careggi, Florence, italy
Locations (1):
- Unit of Clinical Nutrition, University Hospital of Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albanese D, De Filippo C, Cavalieri D, Donati C. Explaining diversity in metagenomic datasets by phylogenetic-based feature weighting. PLoS Comput Biol. 2015 Mar 27;11(3):e1004186. doi: 10.1371/journal.pcbi.1004186. eCollection 2015 Mar. PMID 25815895
- [Background] Borgeraas H, Johnson LK, Skattebu J, Hertel JK, Hjelmesaeth J. Effects of probiotics on body weight, body mass index, fat mass and fat percentage in subjects with overweight or obesity: a systematic review and meta-analysis of randomized controlled trials. Obes Rev. 2018 Feb;19(2):219-232. doi: 10.1111/obr.12626. Epub 2017 Oct 18. PMID 29047207
- [Background] Chung HJ, Yu JG, Lee IA, Liu MJ, Shen YF, Sharma SP, Jamal MA, Yoo JH, Kim HJ, Hong ST. Intestinal removal of free fatty acids from hosts by Lactobacilli for the treatment of obesity. FEBS Open Bio. 2016 Jan 18;6(1):64-76. doi: 10.1002/2211-5463.12024. eCollection 2016 Jan. PMID 27047743
- [Background] Dinan TG, Cryan JF. Melancholic microbes: a link between gut microbiota and depression? Neurogastroenterol Motil. 2013 Sep;25(9):713-9. doi: 10.1111/nmo.12198. PMID 23910373
- [Background] Gomes AC, de Sousa RG, Botelho PB, Gomes TL, Prada PO, Mota JF. The additional effects of a probiotic mix on abdominal adiposity and antioxidant Status: A double-blind, randomized trial. Obesity (Silver Spring). 2017 Jan;25(1):30-38. doi: 10.1002/oby.21671. PMID 28008750
- [Background] Segata N, Izard J, Waldron L, Gevers D, Miropolsky L, Garrett WS, Huttenhower C. Metagenomic biomarker discovery and explanation. Genome Biol. 2011 Jun 24;12(6):R60. doi: 10.1186/gb-2011-12-6-r60. PMID 21702898
- [Background] Verdenelli MC, Ghelfi F, Silvi S, Orpianesi C, Cecchini C, Cresci A. Probiotic properties of Lactobacillus rhamnosus and Lactobacillus paracasei isolated from human faeces. Eur J Nutr. 2009 Sep;48(6):355-63. doi: 10.1007/s00394-009-0021-2. Epub 2009 Apr 14. PMID 19365593
- [Background] John GK, Wang L, Nanavati J, Twose C, Singh R, Mullin G. Dietary Alteration of the Gut Microbiome and Its Impact on Weight and Fat Mass: A Systematic Review and Meta-Analysis. Genes (Basel). 2018 Mar 16;9(3):167. doi: 10.3390/genes9030167. PMID 29547587
- [Background] Sanchez M, Darimont C, Panahi S, Drapeau V, Marette A, Taylor VH, Dore J, Tremblay A. Effects of a Diet-Based Weight-Reducing Program with Probiotic Supplementation on Satiety Efficiency, Eating Behaviour Traits, and Psychosocial Behaviours in Obese Individuals. Nutrients. 2017 Mar 15;9(3):284. doi: 10.3390/nu9030284. PMID 28294985
- [Background] Sanders ME. Probiotics and microbiota composition. BMC Med. 2016 Jun 2;14(1):82. doi: 10.1186/s12916-016-0629-z. PMID 27250499